CLINICAL TRIAL: NCT04921787
Title: Exemplar Hospital Initiation Trial to Enhance Treatment Engagement - Implementation Trial of High Intensity Versus Low Intensity Strategy for Supporting Hospital-Based Opioid Use Disorder Treatment
Brief Title: EXHIT ENTRE Implementation Trial of High Intensity Versus Low Intensity Strategy
Acronym: EXHITENTRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gavin Bart (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Gavin Bart, Gavin Bart, MD PhD FACP DFASAM, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NIDA CTN 0098B; 2UG1DA040316-06 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-06-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; Opioid Use Disorder, Severe; Opioid Use Disorder, Moderate
Keywords: HBOT; MOUD; OUD; SUD; OTP; ED
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Lymphoma, Follicular | interventions — Ultrasonic Waves; Educational Status

STUDY DESIGN:
Intervention Model Description: This is a multi-site, cluster randomized, two group implementation trial comparing a low versus high intensity implementation strategy for supporting hospital-based opioid use disorder treatment (HBOT) in community hospital settings where medication for opioid use disorder (MOUD) treatment has not been implemented. Approximately 24 hospitals meeting defined eligibility requirements, including a desire to address OUD among inpatients through the use of MOUD, will be randomized 1:1 to implement a low- or high-intensity strategy. Hospitals will be randomized with intervention implementation and oversight assigned to one of 3-4 geographically diverse hub academic medical centers with existing clinical and research expertise in HBOT. The randomization will be stratified by site/hub.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity (Active Comparator): MOUD training and support through the use of educational materials.
  Interventions: Other: Low Intensity
- High Intensity (Experimental): MOUD training and support through the use of educational materials in addition to practice facilitation.
  Interventions: Other: High Intensity

INTERVENTIONS:
Other: Low Intensity — Training and education only, a low-intensity strategy inclusive of an HBOT manual, one-time live training on how to use the HBOT manual, and 7 video conference presentations.
  Other Names: Training and education
  Arms: Low Intensity
Other: High Intensity — Practice facilitation, a high-intensity strategy inclusive of low-intensity training, plus practice facilitation that is based in part on a program planning model. This study is a hybrid implementation effectiveness design, testing an implementation strategy while observing and gathering information on the clinical intervention's impact on relevant outcomes.
  Other Names: Practice Facilitation
  Arms: High Intensity

SUMMARY:
This study is a multi-site, cluster randomized, two group implementation trial comparing a low- versus high-intensity implementation strategy for supporting hospital-based opioid use disorder treatment (HBOT) in community hospital settings where medication for opioid use disorder (MOUD) treatment has not been implemented.

DETAILED DESCRIPTION:
The study will randomize approximately 24 community hospitals meeting defined eligibility requirements, including a desire to address OUD among inpatients through the use of MOUD. Community hospitals will be randomized 1:1 to implement a low- or high-intensity strategy. Hospitals will be randomized with intervention implementation and oversight assigned to one of 3-4 geographically diverse hub academic medical centers with existing clinical and research expertise in HBOT. The randomization will be stratified by site/hub. Participants will be assessed for "engagement with MOUD", measured as the proportion of community hospital OUD discharges engaged with MOUD within 34 days following hospital discharge during months 13-24 of the intervention. Further outcomes will be assessed during the entire 4-year study period.

ELIGIBILITY:
Inclusion Criteria:

1. Be a community hospital deemed by the lead investigators to be in the region of a site/hub. Region will usually be defined as state unless a compelling case can be made as to geographic feasibility of implementing the intervention and access to relevant Medicaid data.
2. Be willing to identify a site champion to promote and adopt change that can address OUD in hospitalized patients.
3. Have hospital personnel who state that their institution is interested in and would be willing to work to implement MOUD prior to hospital discharge.
4. Commit to having buprenorphine-waivered prescribers willing and able to write prescriptions to bridge discharged patients to post-discharge OUD treatment, or available direct entry into outpatient MOUD with methadone or buprenorphine.
5. Have hospital staff who express willingness to engage with a site/hub team for training and for data collection.
6. Be willing to be randomized to low-intensity or high-intensity implementation support.
7. Provide inpatient general medical care.
8. Have sufficient numbers of Medicaid OUD discharges (any listed diagnosis; sufficient is defined as at least enough such that when added to the other hospitals in the region there are on average 100 discharges per year). Medicaid data must capture at least 3 discharge diagnoses, outpatient MOUD, and be available within no more than 12 months of discharge.

Exclusion Criteria:

1. Have an ACS routinely prescribing MOUD at discharge.
2. Have an existing, functioning HBOT program or be imminently starting an HBOT initiative, as confirmed by the investigator team.
3. Be a Veterans Affairs hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Engagement with MOUD | 34 days following hospital discharge
  measured as the proportion of community hospital OUD discharges engaged with MOUD within 34 days following hospital discharge during months 13-24 of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Bart, MD,PhD, Principal Investigator — Hennepin Healthcare
Locations (4):
- United States (4):
  - Boston University, Boston, Massachusetts
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - New York University, New York, New York
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Data will be transmitted by the study Data and Statistics Center to the designated party for de-identification, posting, storing, and archiving on the National Institute on Drug Abuse (NIDA) Data Share website. Data Share is an online repository of data from studies funded by the National Institute on Drug Abuse. De-identified individual participant data is expected to be made available.
Supporting Information: Study Protocol
Time Frame: The data will be shared after the primary outcome paper has been accepted for publication, or 18 months after data lock, whichever comes first. The data will remain indefinitely.
Access Criteria: Data from this study will be available to researchers on the website https://datashare.nida.nih.gov/ after the study is complete and the data is analyzed. This website will not include information that can identify individual study participants.The following information will be posted: Study protocol, reference to study publication of primary outcome, data sets (SAS and ASCII ), annotated case report forms, define file (also known as Data Dictionary), study-specific de-identification notes. Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the NIDA Data Share Agreement.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Background] Trowbridge P, Weinstein ZM, Kerensky T, Roy P, Regan D, Samet JH, Walley AY. Addiction consultation services - Linking hospitalized patients to outpatient addiction treatment. J Subst Abuse Treat. 2017 Aug;79:1-5. doi: 10.1016/j.jsat.2017.05.007. Epub 2017 May 11. PMID 28673521
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Derived] Bart G, Korthuis PT, Donohue JM, Hagedorn HJ, Gustafson DH, Bazzi AR, Enns E, McNeely J, Ghitza UE, Magane KM, Baukol P, Vena A, Harris J, Voronca D, Saitz R. Exemplar Hospital initiation trial to Enhance Treatment Engagement (EXHIT ENTRE): protocol for CTN-0098B a randomized implementation study to support hospitals in caring for patients with opioid use disorder. Addict Sci Clin Pract. 2024 Apr 11;19(1):29. doi: 10.1186/s13722-024-00455-9. PMID 38600571